CLINICAL TRIAL: NCT01992484
Title: Association Between the Antiplatelet Drug Efficacy/Safety and Platelet Function in Patients Treated With Novel Platelet Inhibitors Due to an Acute Coronary Syndrome
Brief Title: Platelet Function in Patients With an Acute Coronary Syndrome
Acronym: ATLANTIS-ACS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Jolanta Siller-Matula, PD Dr.med. PhD, Medical University of Vienna
Other Study IDs: ATLANTIS-ACS
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Acute Coronary Syndrome (ACS)
Keywords: platelets, Acute coronary Syndrome (ACS), prasugrel, ticagrelor, aspirin
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aims of the study are to:

* explore whether platelet reactivity in patients treated wih novel platelet inhibitors is associated with clinical outcome
* investigate whether a therapeutic window exist for novel platelet inhibitors
* investigate the incidence of adverse events under treatment with novel platelet inhibitors in the real life clinical scenario
* investigate the association between genetic polymorphisms, inflammation, platelet reactivity and clinical outcome
* investigate synergistic effects between aspirin and novel platelet inhibitors

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Acute coronary syndrome at admission
* Planned treatment with novel platelet inhibitors
* Age >18

Exclusion Criteria:

* Participation in interventional trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with an acute coronary syndrome
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-08; Primary Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Net clinical benefit. | 1 year
  A composite of MACE and BARC=>2 bleedings.

SECONDARY OUTCOMES:
MACE and Major bleeding | 1 year
  MACE: the composite of stent thrombosis, cardiac death and myocardial infarction.
  Major Bleeding: BARC =>2, TIMI major, GUSTO moderate-severe-life threatening.

OTHER OUTCOMES:
single endpoints of acute coronary syndrome, myocardial infarction, cardiac death, all-cause death, urgent vessel revascularization (PCI or CABG), stroke. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Univerity of Vienna, Department of Cardiology, Vienna, Austria